CLINICAL TRIAL: NCT04142346
Title: Postprandial Glucose Responses in Trained Older Adults: Effects of Breaking-up Sedentary Time and 2 Weeks Detraining
Brief Title: Breaking-up Sedentary Time and 2 Weeks Detraining
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lisbon (Other)
Collaborators: Associação Protectora dos Diabéticos de Portugal (Unknown)
Responsible Party: Principal Investigator, Luís Bettencourt Sardinha, Professor, University of Lisbon
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: CEIFMH6/2019
Record Dates: First submitted 2019-10-21; First posted 2019-10-29 (Actual); Last update posted 2019-10-30 (Actual); Status verified 2019-10

CONDITIONS: Old Age
Keywords: sitting time; physical inactivity; breaks; glycemic control; continuous glucose monitoring; older adults
MeSH Terms: conditions — Sedentary Behavior | interventions — Sitting Position

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Uninterrupted sitting (No Intervention): Participants remained seated throughout 7 hours. During the protocol, participants were allowed to go to the bathroom in a wheelchair and al-libitum water was granted.
- Sitting + moderate intensity breaks (Experimental): Participants were instructed to sit throughout 7 hours, while interrupting the sitting position every 30 minutes to perform 2 minutes of moderate-intensity physical activity. The breaks consisted of walk up and down stairs and squats. Each person performed these exercise alternately. During the protocol, participants were allowed to go to the bathroom in a wheelchair and al-libitum water was granted.
  Interventions: Behavioral: Sitting + moderate intensity breaks

INTERVENTIONS:
Behavioral: Sitting + moderate intensity breaks — Participants will be followed in a randomized crossover trial undertaken at Faculty of Human Kinetics between April and August 2019. Participants will attend to the laboratory on twelve separate occasions: visit 1 (day 1), baseline assessments for body composition; visit 2 (day 2), cardiorespiratory fitness assessment; visit 3 (day 3), OGTT and the first randomized experimental protocol; visit 4 (day 4), follow-up OGTT; visit 5 (4-6 days after the first experimental protocol), OGTT and the remaining experimental protocol; visit 6 (day following the previous experimental protocol), follow-up OGTT. An additional 6 visits will be performed following the same rational, after a 2-week period of detraining, where participants will be instructed to refrain from structured exercise. The follow-up assessments for body composition and cardiorespiratory fitness will be accomplished after the protocols.
  Arms: Sitting + moderate intensity breaks

SUMMARY:
Regularly interrupting sedentary behavior (SB) with activity breaks may attenuate postprandial glucose (PPG) excursions and improve glycemic control. The investigators aimed to determine the effect of interrupting 7 hours of prolonged sitting with brief bouts of moderate physical activity (PA) (alternating between up/down stairs and sit/stand up from the chair) on postprandial glucose (PPG) responses in comparison with uninterrupted sitting. In addition, the investigators aimed to examine the effects of 2 weeks of detraining (DT) on PPG on both protocols. Non-diabetic, trained older adults (n = 15) will be recruited for a randomized crossover trial with two treatments performed in two different training conditions: 1) uninterrupted sitting protocol (CON); 2) seated with 2-minutes bouts of moderate PA every 30 minutes (INT). Both protocols will be performed in a trained condition and after 2 weeks of DT. In the early morning of each trial, participants will do an oral glucose tolerance test (OGTT) and 2 blood samples will be collected (fasting and after 2 hours); 2.5 hours after, participants will begin the protocol and two standardized meals will be provided (0 hours and at 3 hours). An iPro2 continuous glucose monitoring (CGM) system will record the average interstitial glucose concentration every 5 minutes. Positive incremental area under the curve (iAUC) and total area under the curve (pAUC) for glucose as well as mean glucose (MG) will be calculated using Matlab. Differences between both protocols and between the two different moments will be examined using generalized estimation equation (GEE), adjusting for sex and age (CI 95%).

DETAILED DESCRIPTION:
Participants will be recruited to take part in a randomized crossover trial using media advertisements and group events within the Lisbon Metropolitan Area. In order to be part of this intervention, the participants will have to be men or women aged between 65 and 90 years-old, physically active, and engaged in structured exercise at least twice a week for the past 6 months. People who have diabetes or any type of physical limitation that would prevent them from performing exercise will be excluded. Power and sample size calculations (G-Power 3.1.9.2) were based on an effect size of 0.78 for the glucose iAUC, a power of 0.80, and a significance of 0.05. The calculation yielded a sample size of 15 participants. This study was approved by the Ethics Committee of the Faculty of Human Kinetics (approval number: 06/2019) and conducted in accordance with the Declaration of Helsinki and with the Convention on Human Rights and Biomedicine. Written informed consents were obtained from all participants.

Participants will be followed in a randomized crossover trial undertaken at Faculty of Human Kinetics between April and August 2019. Participants will attend the laboratory on twelve separate occasions: visit 1 (day 1), baseline assessments for body composition; visit 2 (day 2), cardiorespiratory fitness assessment; visit 3 (day 3), OGTT and the first randomized experimental protocol; visit 4 (day 4), follow-up OGTT; visit 5 (4-6 days after the first experimental protocol), OGTT and the remaining experimental protocol; visit 6 (day following the previous experimental protocol), follow-up OGTT. An additional 6 visits will be performed following the same rational, after a 2-week period of detraining, where participants will be instructed to refrain from structured exercise and reduce their physical activity. The follow-up assessments for body composition and cardiorespiratory fitness will be accomplished after the protocols. Experimental protocol order will be randomized at baseline and on the follow-up period after the detraining process by a third party using a computer-generated list of random numbers (block randomization with balanced block sizes).

On the morning of each intervention day, participants will arrive at the laboratory at 8:00 a.m., after a 10h fast. For 48h prior to intervention day, participants will be asked to refrain from structured moderate-to-vigorous physical activity (MVPA), caffeine and alcohol consumption. Each intervention day will have a total duration of 9.5h and will start with an oral glucose tolerance test. After a baseline blood collection, participants will be instructed to drink an oral glucose drink of 75g dissolved in water (200 ml). Two hours after, another blood sample will be drawn.

At 10:30 a.m., a mixed standard meal (breakfast) will be given to the participants, marking the begging of the 7 hour protocol. The same standard meal will be provided at 1:30 p.m. (lunch). The 200-ml meal will consist of 303 kcal, 42g carbohydrate, 10g fat and 11.2g protein, vitamins and minerals (Nestle Health Science - Resource Energy). The participants will be encouraged to consume the entire meal within 5 minutes. The protocols performed will be: 1) uninterrupted sitting: participants will remain seated throughout 7 hours (SIT); 2) Sitting + moderate intensity breaks: participants will be instructed to sit throughout 7 hours, while interrupting the sitting position every 30 minutes to perform 2 minutes of moderate-intensity physical activity. The breaks will consist of walk up and down the stairs and squats. Each person will perform these exercises alternately. During the protocol, participants will be allowed to go to the bathroom in a wheelchair and al-libitum water will be granted. The following morning after the protocol, the OGTT will be repeated.

ELIGIBILITY:
Inclusion Criteria:

* Men or women
* 65 and 90 years-old
* Physically active
* Engaged in structured exercise at least twice a week for the past 6 months.

Exclusion Criteria:

* Diagnosed with diabetes
* Any type of physical limitation that would prevent them from practicing exercise

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 14 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
Continuous glucose monitoring before and after 2-Weeks of detraining for each intervention protocol (prolonged sitting vs. breaking-up sitting) | 1-month (2 measurement times, one for each protocol, including baseline and after detraining)
  Immediately upon arrival at the laboratory and throughout 24h, a blood glucose monitor (iPro2 CGM with Enlite Sensors MiniMed; Medtronic, Northridge, California, USA) will be placed on the right side of the abdomen. Once inserted, CGM provides interstitial glucose values every 5 minutes. To calibrate the CGM, four capillary blood glucose samples (three in the laboratory and one at home) will be collected and measured using a glucometer (Contour Next One, Ascensia Diabetes Care, Basel, Switzerland).

SECONDARY OUTCOMES:
Postural allocation | 1-month (2 measurement times, one for each protocol, including baseline and after detraining)
  To objectively monitor the experimental protocol, an Activpal (version 5.9.1.1, PAL Technologies, Glasgow, UK) will be attached to the skin on the middle anterior line of the right thigh and will be used continuously during the 7-hour protocol. Data will be collected at a predetermined 10 Hz and in 15 second epochs.
Body Composition | 1-month (2 measurement times (one at baseline and after two weeks of detraining))
  A whole-body scan will be performed and the attenuation of X-rays (DXA) pulsed between 70 and 140 kilovolt synchronously with the line frequency for each pixel of the scanned image that was measured. Abdominal and gynoid body fat mass will be measured through partial analyses of the DXA scan, based on regions of interest (ROIs) set by default on the DXA settings. Following the protocol for DXA described by the manufacturer, a phantom with six fields of acrylic and aluminum of varying thickness and known absorptive properties will be scanned alongside each participant to serve as an external standard for the analyses of different tissue components. The same laboratory technician will position the participants, perform the scans and execute the analyses according to the operator's manual using the standard analysis protocol.
Weight | 1-month (2 measurement times (one at baseline and after two weeks of detraining))
  Participants weight will be measured using an electronic scale with stadiometer (Seca, Hamburg, Germany).
Height | 1-month (2 measurement times (one at baseline and after two weeks of detraining))
  Participants height will be measured using an electronic scale with stadiometer (Seca, Hamburg, Germany).
Cardiorespiratory fitness (CRF) | 1-month (2 measurement times (one at baseline and after two weeks of detraining))
  CRF will be determined using a Modified Bruce Protocol on a motorized treadmill to exhaustion (model Q-65, Quinton, Cardiac Science Corp; Bothell, Washington, USA). All graded tests will be monitored using a 12-lead electrocardiogram. Inspired and expired gases will be continuously analyzed (Quark RMR w/CPET, version 9.1, Cosmed, Rome, Italy). Peak oxygen will be determined as the highest 20 seconds average of the last minute.
Objective Measures of Physical Activity | 1-month (2 measurement times (one week at baseline and during the two weeks of detraining))
  Physical activity will be assessed by accelerometer (ActiGraph, GT3X model, Fort Walton Beach, FL), during participants free living and during the whole two weeks of detraining period. All participants will be asked to wear the device on the right hip. Data will be recorded in 60 second epochs and periods of at least 60 consecutive minutes of zero activity intensity counts will be considered as non-wear time.
Objective Measures of Sedentary Time | 1-month (2 measurement times (one week at baseline and during the two weeks of detraining))
  Sedentary time will be assessed by accelerometer (ActiGraph, CT3X model, Fort Walton Beach, FL), during participants free living and during the whole two weeks of detraining period. All participants will be asked to wear the device on the right hip. Data will be recorded in 60 second epochs and periods of at least 60 consecutive minutes of zero activity intensity counts will be considered as non-wear time.
Upper limb muscle strength | 1-month (2 measurement times (one at baseline and after two weeks of detraining))
  Muscle strength will be assessed on the upper limbs, using the bench press, under isometric conditions (Hyatt, Whitelaw, Bhat, Scott, & Maxwell, 1990; Lovell, Cuneo, & Gass, 2010). The assessment of maximal strength will be performed through a test of isometric supine (multipower, Technogym), with the elbow flexed and the shoulder joint creating an abduction of 90º.
Lower limb muscle strength | 1-month (2 measurement times (one at baseline and after two weeks of detraining))
  Muscle strength will be assessed on the lower limbs, using the leg press machine, under isometric conditions (Hyatt, Whitelaw, Bhat, Scott, & Maxwell, 1990; Lovell, Cuneo, & Gass, 2010). The assessment of the lower limbs will be performed through an isometric test of horizontal Leg Press (S0409, HBP), in which the participant has his thigh flexed and the knee joint creating an angle of 110º.
Phase angle (PhA) | 1-month (2 measurement times (one at baseline and after two weeks of detraining))
  The participants will perform bioimpedence analysis (single frequency, 50 kHz ± 1%, NutriLAB, Akern) in order to determine the PhA. The participants will be in a lying position, with legs apart from each other and arms apart from the trunk, so that the medial surface of the limbs will not touch the rest of the body (Selberg & Selberg, 2002); 4 electrodes (2 in each limb) will be placed on the hand and foot of the dominant side, with a distance of 5 cm between both.
Body Water | 1-month (2 measurement times (one at baseline and after two weeks of detraining))
  The participants will perform bioimpedence analysis (single frequency, 50 kHz ± 1%, NutriLAB, Akern) in order to determine the body water compartments (total body water and extracellular water directly measured and calculated intracellular water). The participants will be in a lying position, with legs apart from each other and arms apart from the trunk, so that the medial surface of the limbs will not touch the rest of the body (Selberg & Selberg, 2002); 4 electrodes (2 in each limb) will be placed on the hand and foot of the dominant side, with a distance of 5 cm between both.
Oral Glucose Tolerance Test | 1-month (4 measurement times, two for each protocol (in the morning of each protocol day and the day after), including baseline and after detraining)
  Baseline blood collection was drawn, and participants were instructed to drink an oral glucose drink of 75g glucose dissolved in water (200ml). Two hours after, another blood sample was collected.

CONTACTS AND LOCATIONS:
Overall Officials: Luis Sardinha, PhD, Principal Investigator — Professor
Locations (1):
- Faculty of Human Kinetics, University of Lisbon, Cruz Quebrada, Portugal